CLINICAL TRIAL: NCT06920901
Title: A Phase 1b, Multicenter, Randomized, Double-blind, Placebo-controlled Study to Evaluate the Safety, Tolerability, Pharmacokinetics, and Immunogenicity of APG777 in Adults With Mild-to-Moderate Asthma
Brief Title: A Study to Evaluate the Safety, Tolerability, Pharmacokinetics (PK), and Immunogenicity of APG777 in Adults With Asthma
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Apogee Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: APG777-105
Record Dates: First submitted 2025-03-27; First posted 2025-04-10 (Actual); Last update posted 2025-09-09 (Actual); Status verified 2025-09

CONDITIONS: Asthma
Keywords: Asthma; Mild to moderate asthma; Tolerability; Immunogenicity; Pharmacokinetics
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- APG777 (Experimental): Participants will receive protocol specified dose of APG7777
  Interventions: Drug: APG777
- Placebo (Placebo Comparator): Participants will receive matching placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: APG777 — APG777 subcutaneous injection
  Arms: APG777
Drug: Placebo — Matching placebo subcutaneous injection
  Arms: Placebo

SUMMARY:
This is a multicenter, randomized, double-blind, placebo-controlled study to evaluate the safety, tolerability, PK, and immunogenicity of APG777 in adult participants with mild-to-moderate asthma.

The duration of the study will be approximately 52 weeks (364 days) for each participant and will consist of a Screening Period, Treatment Period, and Follow-up Period.

ELIGIBILITY:
Inclusion Criteria:

* Have a diagnosis of mild-to-moderate asthma (Global Initiative for Asthma 2023 criteria) ≥ 1 year prior to Screening
* Maintain FeNO-high (≥ 25 parts per billion [ppb]) or FeNO-low (< 25 ppb) status from Screening to Day 1 prior to Randomization
* Pre-bronchodilator forced expiratory volume in 1 second (FEV1) ≥ 60% of predicted normal value at Screening
* Asthma Control Test (ACT) score > 19 at Screening
* Maintained control on as-needed short-acting beta-agonist (SABA) +/- stable dose inhaled corticosteroids (ICS) or stable dose of ICS/ long-acting beta-agonist (LABA); +/- stable dose leukotriene receptor antagonist (LTRA). ICS dose should be stable for ≥ 12 weeks prior to Day 1, LTRA dose should be stable for ≥ 8 weeks prior to Day 1
* Women of childbearing potential and male participants to use a highly effective form of contraception

Exclusion Criteria:

* Any asthma exacerbation requiring systemic corticosteroids within 12 weeks of Screening and/or any asthma exacerbation that resulted in overnight hospitalization within 6 months prior to Screening
* Any history of life-threatening asthma, defined as an asthma episode that required intubation and/or was associated with hypercapnia
* History of biologics use for treatment or control of asthma
* Current smokers or participants with a smoking history of ≥ 10 pack years
* Known history of illicit drug abuse, harmful alcohol use

Note: Other protocol defined criteria may apply.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2025-03-27 (Actual); Primary Completion 2026-09 (Estimated); Study Completion 2027-03 (Estimated)

PRIMARY OUTCOMES:
Number of Participants with Treatment Emergent Adverse Events (TEAEs) | Up to 52 weeks
Number of Participants with Abnormal Laboratory Findings | Up to 52 weeks
Number of Participants with Abnormal Vital Signs | Up to 52 weeks
Number of Participants with Abnormal Electrocardiograms (ECGs) | Up to 52 weeks
Number of Participants with Abnormal Physical Examination Findings | Up to 52 weeks

SECONDARY OUTCOMES:
Maximum concentration (Cmax) of APG777 | Up to 48 weeks
Time to reach Cmax (tmax) | Up to 48 weeks
Terminal elimination rate constant (λz) | Up to 48 weeks
Terminal Elimination half-life (t1/2) | Up to 48 weeks
Area Under the Serum Concentration-time curve (AUC) from Time 0 to the Last Quantifiable Time Point (AUC0-last) | Up to 48 weeks
AUC From Time 0 Extrapolated to Infinity (AUC0-inf) | Up to 48 weeks
Apparent Clearance of APG777 (CL/F) | Up to 48 weeks
Apparent Volume of Distribution (Vz/F) | Up to 48 weeks
Number of Participants with Anti-Drug-Antibodies (ADAs) | Up to 48 weeks
Cmax in Participants With and without ADAs | Up to 48 weeks
AUClast Participants With and without ADAs | Up to 48 weeks
AUCInf Participants With and without ADAs | Up to 48 weeks

CONTACTS AND LOCATIONS:
Locations (11):
- United States (9):
  - Investigational Site, La Jolla, California
  - Investigational Site, Long Beach, California
  - Investigational Site, San Jose, California
  - Investigational Site, Torrance, California
  - Investigational Site, Normal, Illinois
  - Investigational Site, Kansas City, Missouri
  - Investigational Site, Edmond, Oklahoma
  - Investigational Site, Philadelphia, Pennsylvania
  - Investigational Site, Pittsburgh, Pennsylvania
- United Kingdom (2):
  - Investigational Site, Bradford, West Yorkshire
  - Investigational Site, Manchester